CLINICAL TRIAL: NCT04403126
Title: Implementation of Forgiveness Education to Increase Psychological Well-being in Three Culturally Distinct Areas: Northern Ireland, Israel/Palestine, and Taiwan
Brief Title: To Increase Psychological Well-being by the Implementation of Forgiveness Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Stranmillis University College, Northern Ireland (Unknown); Hebrew University of Jerusalem (Other); National Chung Cheng University, Taiwan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-0432; EDUC/EDUC PSYCH (Other: University of Wisconsin); A173000 (Other: University of Wisconsin)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Anger; Depressive Symptoms; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Classrooms participating in this study will be randomly assigned to either an experimental group (with forgiveness intervention) or a control group (with regular instruction). The experimental group will receive the 1st forgiveness intervention for 12 weeks and then the control group will turn into an experimental group to receive a 2nd forgiveness intervention for 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forgiveness curriculum for 5th grade (Experimental): Classrooms randomly assigned to the experimental group will receive the forgiveness intervention. The forgiveness intervention will follow the curriculum - "The Journey Toward Forgiveness -A Guided Curriculum for Children Ages 10-12 (Grade 5 in the US)". The Forgiveness Curriculum Guide consists 14 lessons over 12 weeks. Each class meets weekly for 40 to 60 minutes to complete one lesson (in two of the weeks, there will be two lessons).
  Interventions: Other: forgiveness education intervention
- Regular school instruction (No Intervention): Classrooms randomly assigned to the control group will have instruction as usual.

INTERVENTIONS:
Other: forgiveness education intervention — The forgiveness education intervention primarily teaches the concept of forgiveness through stories. We chose the kind of stories that should appeal to children ages 10 through 12. Each lesson is planned according to the following procedure: story-telling/movie-watching, discussion, and in-class activities.
  Arms: Forgiveness curriculum for 5th grade

SUMMARY:
This project examines the development of psychological well-being in children and teachers through a 12- week forgiveness education program conducted in three conflict zones of the world, Northern Ireland, Israel/Palestine, and Taiwan.

A 12-week forgiveness education program will be investigated in elementary schools in three conflict zones of the world, Northern Ireland, Israel/Palestine, and Taiwan. The responsibilities of the sub-team in each of the three research sites will be:

* a. recruiting schools, assisting the teacher training before the forgiveness education program starts
* b. shepherding teachers, doing the fidelity checks, administering the instruments and collecting data during the forgiveness education program.

Once a school gives permission to be part of this study, the forgiveness curriculum will be implemented as a 12-week standard curriculum for the grade 5 (US equivalency) students. Teachers of the grade 5 classes will be trained to administer the program. Teachers, students and their parents must give the consent to take part in the measures of the study.

DETAILED DESCRIPTION:
Classrooms participating in this study will be randomly assigned to either an experimental or a control group. The experimental group will receive the 1st forgiveness intervention for 12 weeks and then the control group will turn into an experimental group to receive a 2nd forgiveness intervention for 12 weeks.

In order to assess if such education increases psychological well-being in students (children) and teachers (adults), teachers and students in both groups will receive the same measures for four times in the study: within one week before the 1st forgiveness intervention, within one week after the 1st forgiveness intervention, within one week after the 2nd forgiveness intervention, four weeks after the 2nd forgiveness intervention.

The instruments include: for teachers, the assessment data will consist of the Enright Forgiveness Inventory Short Form (EFI-30), the Patient-Reported Outcomes Measurement Information System (PROMIS): Anger, Anxiety, and Depression scales, the Ethnic Prejudice Scale, the Herth Hope Index, the Rosenberg Self-Esteem Scale, a Classroom Cooperation scale, and a Cross-Cultural Exit Interview (written questionnaire). For students, the assessment data will consist of the Enright Forgiveness Inventory for Children (EFI-C), the PROMIS measures for pediatric self-report (ages 8-17): Anger, Anxiety, and Depressive Symptoms scales, the Ethnic Prejudice Scale for children, the Children's Hope Scale, the Coopersmith Self-Esteem Inventory (School Form), and academic achievement (likely to be scores/grades of Math, writing and reading in their own language). After the 2nd forgiveness intervention, select participants (teachers and children) will take part in individual interviews.

ELIGIBILITY:
Inclusion Criteria:

* Students in 5th grade (US equivalency, aged 10-12)
* Teachers in 5th grade (US equivalency)

Exclusion Criteria:

* Students who are in grades other than 5th grade
* Teachers who are in grades other than 5th grade

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1300 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in forgiveness in adult (teachers) after forgiveness intervention assessed by EFI-30. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  Enright Forgiveness Inventory Short Form (EFI-30), scores range from 30 to 180 with higher scores representing higher levels of forgiveness, which is a better outcome.
Change in forgiveness in child (students) after forgiveness intervention assessed by EFI-C. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  Enright Forgiveness Inventory for Children (EFI-C): scores range from 30 to 120 with higher scores representing higher levels of forgiveness, which is a better outcome.
Change in anger in adult (teachers) after forgiveness intervention assessed by PROMIS Measures. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Patient Reported Outcome Measurement Information System (PROMIS) Anger Short Form: scores range from 5 to 25 with higher scores representing higher levels of anger, which is a worse outcome.
Change in anger in child (students) after forgiveness intervention assessed by PROMIS Measures. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Patient Reported Outcome Measurement Information System (PROMIS) Measures for Pediatric (ages 8-17) Anger Short Form: scores range from 5 to 25 with higher scores representing higher levels of anger, which is a worse outcome.
Change in anxiety in adult (teachers) after forgiveness intervention assessed by PROMIS Measures. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Patient Reported Outcome Measurement Information System (PROMIS) Anxiety Short Form: scores range from 5 to 40 with higher scores representing higher levels of anxiety, which is a worse outcome.
Change in anxiety in child (students) after forgiveness intervention assessed by PROMIS Measures. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Patient Reported Outcome Measurement Information System (PROMIS) Measures for Pediatric (ages 8-17) Anxiety Short Form: scores range from 5 to 40 with higher scores representing higher levels of anxiety, which is a worse outcome.
Change in depression in adult (teachers) after forgiveness intervention assessed by PROMIS Measures. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Patient Reported Outcome Measurement Information System (PROMIS) Depression Short Form, scores range from 5 to 40 with higher scores representing higher levels of depression, which is a worse outcome.
Change in depression in child (students) after forgiveness intervention assessed by PROMIS Measures. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Patient Reported Outcome Measurement Information System (PROMIS) Measures for Pediatric (ages 8-17) Depressive Symptoms Short Form: scores range from 5 to 40 with higher scores representing higher levels of depression, which is a worse outcome.
Change in prejudice in adult (teachers) after forgiveness intervention assessed by the Ethnic Prejudice Scales. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Ethnic Prejudice Scale: scores range from 20 to 100 with higher scores representing higher levels of prejudice, which is a worse outcome.
Change in prejudice in child (students) after forgiveness intervention assessed by the Ethnic Prejudice Scales. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  Ethnic Prejudice Scales: wording changes in the adult form of the Ethnic Prejudice Scale will be made to bring it to the level of 5th grade students (aged 10-12). Scores range from 20 to 100 with higher scores representing higher levels of prejudice, which is a worse outcome.
Change in hope in adult (teachers) after forgiveness intervention assessed by Herth Hope Index. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  Herth Hope Index: scores range from 12 to 48 with higher scores representing more hopefulness, which is a better outcome.
Change in hope in child (students) after forgiveness intervention assessed by Children's Hope Scale. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Children's Hope Scale: scores range from 6 to 36with higher scores representing more hopefulness, which is a better outcome.
Change in self-esteem in adult (teachers) after forgiveness intervention assessed by the Rosenberg Self-Esteem Scale. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Rosenberg Self-Esteem Scale: scores range from 10 to 40 with higher scores representing higher self-esteem, which is a better outcome.
Change in self-esteem in child (students) after forgiveness intervention assessed by the Coopersmith Self-Esteem Inventory. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  Coopersmith Self-Esteem Inventory Short Form: scores range from 0 to 25 with higher scores representing higher self-esteem, which is a better outcome.
Change in classroom cooperation in students after forgiveness intervention assessed by the Classroom Cooperation Scale. | Baseline, up to 14 weeks, up to 31 weeks, up to 34 weeks.
  The Classroom Cooperation Scale is teachers' measure of student cooperation, scores range from 10 to 40 with higher scores representing higher level of cooperation, which is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Enright, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD will be shared beginning 1 year and ending 5 years following the first article publication, with anyone who wished to access the data for any purpose.
Access Criteria: Data requestors will need to contact renright@wisc.edu to gain access to the data. Data are available for 5 years at a third party website (Link to be included).

REFERENCES:
- [Background] Akhtar S, Barlow J. Forgiveness Therapy for the Promotion of Mental Well-Being: A Systematic Review and Meta-Analysis. Trauma Violence Abuse. 2018 Jan;19(1):107-122. doi: 10.1177/1524838016637079. Epub 2016 Mar 23. PMID 27009829
- [Background] Wade NG, Hoyt WT, Kidwell JE, Worthington EL. Efficacy of psychotherapeutic interventions to promote forgiveness: a meta-analysis. J Consult Clin Psychol. 2014 Feb;82(1):154-70. doi: 10.1037/a0035268. Epub 2013 Dec 23. PMID 24364794
- [Background] Reed GL, Enright RD. The effects of forgiveness therapy on depression, anxiety, and posttraumatic stress for women after spousal emotional abuse. J Consult Clin Psychol. 2006 Oct;74(5):920-9. doi: 10.1037/0022-006X.74.5.920. PMID 17032096
- [Background] Baxter SD, Smith AF, Litaker MS, Baglio ML, Guinn CH, Shaffer NM. Children's Social Desirability and Dietary Reports. J Nutr Educ Behav. 2004 Mar-Apr;36(2):84-9. doi: 10.1016/s1499-4046(06)60138-3. PMID 15068757
- [Background] Snyder CR, Hoza B, Pelham WE, Rapoff M, Ware L, Danovsky M, Highberger L, Rubinstein H, Stahl KJ. The development and validation of the Children's Hope Scale. J Pediatr Psychol. 1997 Jun;22(3):399-421. doi: 10.1093/jpepsy/22.3.399. PMID 9212556
- [Background] Freedman SR, Enright RD. Forgiveness as an intervention goal with incest survivors. J Consult Clin Psychol. 1996 Oct;64(5):983-92. doi: 10.1037//0022-006x.64.5.983. PMID 8916627
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Enright RD, Santos MJ, Al-Mabuk R. The adolescent as forgiver. J Adolesc. 1989 Mar;12(1):95-110. doi: 10.1016/0140-1971(89)90092-4. PMID 2708604
- [Background] Cattell RB. The Scree Test For The Number Of Factors. Multivariate Behav Res. 1966 Apr 1;1(2):245-76. doi: 10.1207/s15327906mbr0102_10. No abstract available. PMID 26828106
- [Background] CRANDALL VC, CRANDALL VJ, KATKOVSKY W. A CHILDREN'S SOCIAL DESIRABILITY QUESTIONNAIRE. J Consult Psychol. 1965 Feb;29:27-36. doi: 10.1037/h0020966. No abstract available. PMID 14277395
- [Background] CROWNE DP, MARLOWE D. A new scale of social desirability independent of psychopathology. J Consult Psychol. 1960 Aug;24:349-54. doi: 10.1037/h0047358. No abstract available. PMID 13813058
- [Background] HORN JL. A RATIONALE AND TEST FOR THE NUMBER OF FACTORS IN FACTOR ANALYSIS. Psychometrika. 1965 Jun;30:179-85. doi: 10.1007/BF02289447. No abstract available. PMID 14306381